CLINICAL TRIAL: NCT05344573
Title: Optimizing Pulsatility During Cardiopulmonary Bypass to Reduce Acute Kidney Injury: Prospective Observational Study
Brief Title: Optimizing Pulsatility During Cardiopulmonary Bypass
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-2465; K23HL151882 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-04-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Endothelial Dysfunction; Acute Kidney Injury
Keywords: Endothelial function; Acute Kidney Injury; Cardiopulmonary bypass; Cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Vascular tissue Bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-pulsatile cardiopulmonary bypass: Subjects who undergo cardiac surgery with non-pulsatile cardiopulmonary bypass
- Pulsatile cardiopulmonary bypass: Subjects who undergo cardiac surgery with pulsatile cardiopulmonary bypass

SUMMARY:
Cardiopulmonary bypass during cardiac surgery provides blood flow to the body during surgery but has adverse effects on different organs. Blood flow during cardiopulmonary bypass may be pulsatile or non-pulsatile, which may impact normal organ function after surgery. The study will collect data on the type of cardiopulmonary bypass used during surgery and organ function to determine if there is an association between the type of bypass and organ function.

DETAILED DESCRIPTION:
Cardiac surgery is a high-risk elective surgical procedure frequently requiring CPB in which a machine pumps blood while the surgeon operates on the heart. CPB contributes to surgical risk by causing endothelial dysfunction and acute kidney injury (AKI). Endothelial dysfunction and AKI happen because heart lung machines typically generate non-pulsatile blood flow, which is abnormal and results in impaired tissue oxygen delivery. Normal blood flow is pulsatile due intermittent contraction and relaxation of the heart during the cardiac cycle, which produces a mechanical signal that induces endothelial cells to produce nitric oxide. Without nitric oxide, blood flow does not penetrate as deeply into organs such as the kidneys which leads to acute kidney injury. AKI increases mortality 10-fold after cardiac surgery placing many people at risk since over 400,000 people have surgery with CPB each year in the United States. Thus, pulsatile CPB may influence endothelial function and renal blood flow after cardiac surgery. This study will observe patients undergoing cardiac surgery with CPB and compare patients who receive pulsatile or non-pulsatile CPB.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 70
* Able to provide informed consent
* Scheduled for elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Patients undergoing emergency procedures
* Diagnosed with sepsis
* Experiencing delirium
* Experiencing hemodynamic instability (heart rate > 100 and systolic blood pressure < 90)
* Patients with a mechanical circulatory support device
* Requiring vasoactive medications before surgery
* Patients with a reduced left ventricular ejection fraction (less than 50%)
* Patients with a contraindication to transesophageal echocardiography

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 50 to 70 years scheduled for elective cardiac surgery with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Percent change in flow mediated dilation of the brachial artery after cardiac surgery

SECONDARY OUTCOMES:
Acute kidney injury | From intensive care unit admission after surgery to intensive care unit discharge, up to 7 days
  Acute kidney injury by the KDIGO criteria
Renal blood flow velocity | Intra-operative time point: after cardiopulmonary bypass, up to 12 hours
  Renal blood flow velocity measured by pulse wave doppler
Acute kidney injury risk | Measured 4 hours after the end of cardiopulmonary bypass, up to 12 hours
  Acute kidney injury risk measured by urinary TIMP2*IGFBP7
Perioperative death | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Death after surgery during the surgical hospital encounter
Myocardial infarction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Myocardial infarction after surgery
Stroke | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Stroke after surgery
New renal failure requiring renal replacement therapy | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New renal failure requiring renal replacement therapy after surgery
Re-exploration for bleeding | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Need for surgical re-exploration to control hemorrhage
Post-operative sepsis | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative sepsis determined by positive blood culture
New onset atrial fibrillation | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative new onset atrial fibrillation
Post-operative blood loss | From intensive care unit admission to 24 hours after intensive care unit admission, up to 24 hours
  Post-operative blood loss determined by total surgical drain output
Duration of mechanical ventilation | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Duration of mechanical ventilation after surgery
Post-operative delirium | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative delirium determined by the Confusion Assessment Method for the Intensive Care Unit score
Post-operative hospital length of stay | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Duration of hospital stay after surgery
New requirement for mechanical circulatory support | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative initiation of mechanical circulatory support
Intra-operative red blood cell transfusion | During the intra-operative time period, up to 12 hours
  Intra-operative red blood cell transfusion in units
Post-operative red blood cell transfusion | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative red blood cell transfusion in units
Post-operative platelet transfusion | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative platelet transfusion in units
Post-operative plasma transfusion | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative plasma transfusion in units
Post-operative cryoprecipitate transfusion | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative cryoprecipitate transfusion in units
Intra-operative platelet transfusion | During the intra-operative time period, up to 12 hours
  Intra-operative platelet transfusion in units
Intra-operative plasma transfusion | During the intra-operative time period, up to 12 hours
  Intra-operative plasma transfusion in units
Intra-operative cryoprecipitate transfusion | During the intra-operative time period, up to 12 hours
  Intra-operative cryoprecipitate transfusion in units
Glycocalyx thickness | Start of the intra-operative period to 24 hours after intensive care unit admission
  Glycocalyx thickness determined by sublingual microcirculation microscopy
Microvascular circulatory function | Start of the intra-operative period to 24 hours after intensive care unit admission
  Microvascular circulatory function determined by sublingual microcirculation microscopy
New onset of acute lung injury | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Diagnosis of acute lung injury by PaO2 to FiO2 ratio
New onset of left ventricular diastolic dysfunction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Diagnosis new onset diastolic dysfunction by annular e' velocity: septal e' < 7 cm/sec, lateral e' <10 cm/sec, average E/e' ratio > 14, LA volume index > 34 mL/m2, and peak TR velocity > 2.8 m/sec.
New onset of left ventricular systolic dysfunction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New onset of left ventricular systolic dysfunction determined by a LV ejection fraction <50%
New onset of right ventricular systolic dysfunction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New onset of right ventricular systolic dysfunction determined by a tricuspid annular plane systolic excursion less than 16 mm

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Clendenen, MD, MS, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No